CLINICAL TRIAL: NCT05733559
Title: An Observational Prospective Clinical Study to Assess Clinical Performance of QIAstat-Dx® Respiratory Panel Plus (RPP) SARS-CoV-2 Target in the Intended Use Population and Environment
Brief Title: QIAstat-Dx® Respiratory Panel Plus (RPP) Clinical Performance Study
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: DHF-18-0127-0-CSP-003
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-10

CONDITIONS: Respiratory Disease
Keywords: Respiratory Virus; SARS-CoV-2 coronavirus
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal Swab (NPS) collected per the manufacturer's instructions and eluted in Universal Transport Media (UTM) from subjects with signs and symptoms of respiratory infection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: QIAstat-Dx® Respiratory Panel Plus (RPP) — An observational prospective performance evaluation study of QIAstat-Dx® Respiratory Panel Plus (RPP) SARS-CoV-2 target against a marketed comparator, using NPS collected per the manufacturer's instructions and eluted in Universal Transport Media (UTM) from subjects with signs and symptoms of respiratory infection

SUMMARY:
This study will evaluate the clinical performance of the QIAstat-Dx® Respiratory Panel Plus (RPP) SARS-CoV-2 target with a validated comparator method

DETAILED DESCRIPTION:
This multicentre study aims to evaluation the clinical performance of the QIAstat-Dx® Respiratory Panel Plus (RPP) SARS-CoV-2 target with a validated comparator method

ELIGIBILITY:
Inclusion Criteria:

* Presenting with signs and symptoms of a respiratory infection.
* Consent or assent to be obtained
* Able to communicate (speak, read and write) in local language, and able to understand and sign the required study documents.
* Willing and able to provide Nasopharyngeal Swab (NPS) Specimen collected per manufacturer's instructions.

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, are unsuitable for participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptoms of respiratory infection
Sampling Method: Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
PPA | 8 weeks
  positive percentage agreement
NPA | 8 weeks
  negative percentage agreement

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Study Director — QIAGEN Gaithersburg, Inc
Locations (1):
- QIAGEN, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No